CLINICAL TRIAL: NCT01208077
Title: PROGNOSTIC HEMODYNAMIC PROFILING IN THE ACUTELY ILL EMERGENCY DEPARTMENT PATIENT
Brief Title: PREMIUM Registry: PRognostic HEModynamIc Profiling in the AcUtely Ill EMergency Department Patient
Acronym: PREMIUM
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Collaborators: BMEYE BV the Netherlands (Unknown); Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Richard M Nowak, Sr, Staff Emergency Medicine, Henry Ford Health System
Other Study IDs: Protocol: HFH DEM 002
Record Dates: First submitted 2010-09-14; First posted 2010-09-23 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2015-08

CONDITIONS: Acute CHF; Acute Stroke Syndromes; Systemic Infections
Keywords: ED hemodynamic profiles; patients treated under current clinical standards; Acute CHF; Stroke syndromes; Systemic infection
MeSH Terms: conditions — Toxemia; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute CHF: 1. Recurrent or worsening (within 3 days) shortness of breath as the primary presenting ED complaint
  2. Initial treating ED physician impression that the worsening dyspnea is most likely caused by decompensated CHF
  3. Known history of physician diagnosed CHF
  4. Natriuretic peptide (BNP, MR-pro ANP, NT pro BNP) level will be ordered by the treating physician as part of the patient's work up
- Acute Stroke Syndrome: 1. Onset of abnormal neurological symptoms consistent with possible stroke, within the prior 24 hours, as the primary ED complaint
  2. Initial treating ED physician impression that the abnormal neurological symptoms/signs are most likely caused by an acute stroke syndrome
  3. Non contrast head CT will be ordered by the treating physician as part of the patient's work up
- Acute Systemic Infection: 1. Any combinations of acute (within 3 days) symptoms and signs that the treating ED physician, after initial history and physical examination, attributes to a systemic infection
  2. Blood cultures and/or a blood lactate will be ordered by the treating physician as part of the patient's work up

SUMMARY:
This multinational registry (3 USA, 2 European centers) will capture in the ED continuous non invasive hemodynamic monitoring (using Nexfin finger cuff technology) of patients presenting with acute heart failure, stroke syndromes and systemic infection. Patients will be observed after their Emergency Department (ED) disposition to determine clinical outcomes (length of stay in the hospital, the development of any organ dysfunction, mortality and need for unscheduled medical care within the ensuing 30 days). It is anticipated that specific ED hemodynamic profiles will be predictive of better clinical outcomes than others. This information will provide the outcome data needed to design future therapeutic trials that will evaluate the effect of ED hemodynamic manipulations on overall patient management and outcomes.

DETAILED DESCRIPTION:
The PREMIUM Registry is a multinational, prospective, observational convenience study of the ED hemodynamic profiles of patients presenting with acute CHF, stroke and systemic infections and their potential relationship with patient outcomes. Continuous hemodynamics will be measured by noninvasive means using the Nexfin device and outcomes (in hospital length of stay, the interval development of organ dysfunction and mortality or the need for unscheduled medical care within the ensuing 30 days) will be captured within the registry.

The treating ED physicians will be blinded to the hemodynamic monitoring and there will be no modification of the standard care that each patient receives. Hospital charts will be reviewed and patients/family members will be additionally called at 30 days after the hospital visit in order to collect any additional outcome data.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* 18 years of age or older
* Able to provide informed consent
* No initiated therapy since arrival to the ED
* Must be enrolled within 4 hours of arrival to the ED

Inclusion Criteria for Acute CHF

* Recurrent or worsening (within 3 days) shortness of breath as the primary presenting ED complaint
* Initial treating ED physician impression that the worsening dyspnea is most likely caused by decompensated CHF
* Known history of physician diagnosed CHF
* Natriuretic peptide (BNP, MR-pro ANP, NT pro BNP) level will be ordered by the treating physician as part of the patient's work up

Inclusion Criteria for Acute Stroke Syndrome

* Onset of abnormal neurological symptoms consistent with possible stroke, within the prior 24 hours, as the primary ED complaint
* Initial treating ED physician impression that the abnormal neurological symptoms/signs are most likely caused by an acute stroke syndrome
* Non contrast head CT will be ordered by the treating physician as part of the patient's work up

Inclusion Criteria for Acute Systemic Infection

* Any combinations of acute (within 3 days) symptoms and signs that the treating ED physician, after initial history and physical examination, attributes to a systemic infection
* Blood cultures and/or a blood lactate will be ordered by the treating physician as part of the patient's work up

Exclusion Criteria:

General Exclusion Criteria

* ESRD requiring hemo or peritoneal dialysis
* Suspected pregnancy
* Not able to be followed up in 30 days
* Patients with "comfort only" DNR status
* Patients with known STEMI
* Excessive agitation
* Transferred from another treating facility
* Known aortic valve disease
* On continuous IV home infusions (such as milrinone, primacor)
* Known Left Ventricular Assist device (LVAD)
* Known prior enrollment in this study
* In current therapeutic Investigational study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be screened and enrolled from the Emergency Department
Sampling Method: Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2010-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Hemodynamic profile (CO, SVR, SV, DP/DT and Indexed values) | 4 hours
  Describe the 4 hour continuous ED hemodynamic profiles (CO, SVR, SV, DP/DT and Indexed values)of patients treated under current clinical standards with acute CHF, stroke syndromes and systemic infection.

SECONDARY OUTCOMES:
Hemodynamic Profiles in acute CHF, stroke, and systemic infection | 4 Hours
  Describe the hemodynamic profiles within existing risk stratification groupings currently used for these 3 disease states. These include but are not limited to BNP and troponin values for acute CHF, infarct/bleed size in acute stroke syndromes, and WBC and procalcitonin (where applicable) and blood lactate levels in systemic infections.
  Determine which hemodynamic profiles measured in the ED predict clinical outcomes (mortality, end organ dysfunction, and length of stay)

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Nowak, MD, Principal Investigator — Henry Ford Health System
Locations (4):
- United States (2):
  - Detroit Receiving Hospital/Wayne State University, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
- University LaSapienza Rome Sant'Andrea Hospital, Rome, Rome, Italy
- VU University Medical Centre, Amsterdam, Amsterdam, Netherlands